CLINICAL TRIAL: NCT05256238
Title: Improving Health-related Quality of Life of Head and Neck Cancer Patients Via a Dedicated Comprehensive Supervised Exercise Program (CSEP)
Brief Title: Effect of Exercise in Head and Neck Cancer Patients
Acronym: EffEx-HN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Kom Op Tegen Kanker (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: s65549
Record Dates: First submitted 2021-11-23; First posted 2022-02-25 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Cancer
Keywords: exercise program
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- usual supportive care + comprehensive supervised exercise program (CSEP) (Experimental)
  Interventions: Other: comprehensive supervised exercise program (CSEP)
- usual supportive care (No Intervention)

INTERVENTIONS:
Other: comprehensive supervised exercise program (CSEP) — The CSEP starts as soon as possible after cancer diagnosis and lasts for 12 weeks:
  * week 1-6 (during cancer treatment): 2 supervised sessions at the exercise room of the University Hospital Leuven in connection to the radiotherapy treatment session and one additional session at home. Patients will receive equipment to perform the program at home, e.g. weights, therabands,…
  * week 7-12 (after cancer treatment): 1 supervised session at the exercise room of University Hospital Leuven in connection to the follow-up consultations (once a week) with the oncologist and two additional sessions at home
  * maintenance program (from week 13), patients will exercise at home with a monthly teleconsultation
  Arms: usual supportive care + comprehensive supervised exercise program (CSEP)

SUMMARY:
Head and neck cancers (HNC) are malignancies originating from the mucosa in the oral cavity, nasopharynx, oropharynx, hypopharynx and larynx. Unfortunately, the majority of patients with HNC have locally advanced disease at diagnosis and should, therefore, be treated with chemoradiotherapy (CRT) or with radical surgery followed by adjuvant (C)RT. Treatment of HNCs with (C)RT frequently results in serious and persistent impairments in physical and psychosocial functioning. In order to prevent worsening of a person's functioning at diagnoses and limit the physical impact of the treatments for HNC, a comprehensive supervised exercise program (CSEP) is needed early during treatment.

There is a need to improve integration of exercise programs into HNC care with aim to help head and neck cancer patients regain physical, mental and social functioning. Currently, no program is available adapted to the specific needs of head and neck cancer patients, in particular during cancer treatment.

The primary scientific objective is to examine the effectiveness of a comprehensive supervised exercise program, in addition to usual care, on health-related quality of life (primary outcome parameters) during treatment of head and neck cancer, compared to usual care only, up to 1 year after diagnosis.

Secondary objectives entail gathering information on the effectiveness of the CSEP, in addition to usual care on secondary outcome parameter such as physical and mental functioning, activity level and participation level; to determine the feasibility of such CSEP (defined as at least 50% of eligible patients enrolling in the study and completing at least 50% of the planned intervention sessions) and possible barriers and facilitators for participating in a CSEP during head and neck cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Diagnosed with primary malignant tumour head and neck region (oral cavity, nasal cavity and paranasal sinuses, pharynx, larynx, salivary glands, thyroid)
* ECOG performance score 0-1
* Planned for curative (chemo)radiotherapy
* Able to complete baseline assessments prior to start of radiotherapy.
* Physically and mentally capable of taking part in an exercise program and motivated to engage in a supervised exercise program.

Exclusion Criteria:

* Patients < 18 years
* ECOG ≥ 2
* Patient with HNC, treated with palliative intent
* Evidence of distant metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | 6 months post-diagnosis
  Health-related quality of life will be measured with the European Organisation for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.

SECONDARY OUTCOMES:
Health-related quality of life: physical functioning | 6 months
  The physical functioning subscale of the European Organisation for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30) 6 months post-diagnosis is the key secondary outcome.
Disease-specific health-related quality of life | baseline- 6 weeks -12 weeks- 6 months - 12 months post-diagnosis
  Disease-specific health-related quality of life will be measured with the revised European Organisation for Research and Treatment of Cancer Head and Neck Cancer Module (EORTC-QLQ-HN43). EORTC QLQ-HN43 module has 43 questions and is combined into 12 scales (Fear of Progression, Body Image, Dry Mouth and Sticky Saliva, Pain in the Mouth, Sexuality, Problems with Senses, Problems with Shoulder, Skin Problems, Social Eating, Speech, Swallowing and Problems with Teeth) and 7 single items (Coughing, Swelling in the Neck, Neurological Problems, Trismus, Social Contact, Weight Loss and Wound Healing). All of the scales and single-item measures range in score from 0 to 100. For all items and scales, high scores indicate more problems.
Physical function: Pain | baseline- 6 weeks -12 weeks- 6 months - 12 months post-diagnosis
  Pain will be measured using the Brief Pain Inventory (questionnaire), a self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. The patient is asked to rate their worst, least, average, and current pain intensity, list current treatments and their perceived effectiveness, and rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a 10 point scale.
Physical function: Fatigue | baseline- 6 weeks -12 weeks- 6 months - 12 months post-diagnosis
  The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) is a 40-item measure that assesses self-reported fatigue and its impact upon daily activities and function (questionnaire). FACIT-F scores range between 0 and 52, with higher scores indicating less fatigue.
Upper limb strength | baseline- 6 weeks -12 weeks- 6 months - 12 months post-diagnosis
  A Jamar handheld dynamometer will be used to measure upper limb strength.
Lymphedema: neck circumference measurement | baseline- 6 weeks -12 weeks- 6 months - 12 months post-diagnosis
  The presence of lymphedema will be evaluated with tape measurement of the neck circumference
Lymphedema: %water content | baseline- 6 weeks -12 weeks- 6 months - 12 months post-diagnosis
  %water content will be measured with the MoisturemeterD Compact (tissue dielectric constant (TDC) measurement)
Lymphedema: self-reported | baseline- 6 weeks -12 weeks- 6 months - 12 months post-diagnosis
  Self-reported lymphedema will be assessed with the Lymphedema Symptom Intensity and Distress Survey - Truncal and Head and Neck (LSIDS-H&N).This tool was developed specifically to measure lymphedema symptoms in HNC patients. The tool asks participants to indicate the presence of a symptom (yes or no). Participants then rate all yes symptoms for intensity and distress on two separate 10-point numeric scales.
Shoulder forward flexion and abduction range of motion | baseline- 6 weeks -12 weeks- 6 months - 12 months post-diagnosis
  The range of motion of both shoulder forward flexion and abduction will be measured using an inclinometer
Physical fitness | baseline- 6 weeks -12 weeks- 6 months - 12 months post-diagnosis
  The 6 minute walking distance (6MWD) will be used to evaluate physical fitness. This is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome.
Body composition: amount of fat, bone, water, and muscle in the body | baseline- 6 weeks -12 weeks- 6 months - 12 months post-diagnosis
  Body composition will be assessed through Bio-impedance Spectroscopy with InBody device. Bioelectrical Impedance Analysis (BIA) is a method of quantifying body composition by introducing an electrical current throughout the body. InBody uses this method to measure body composition, which divides the persons weight into different components, such as water, lean body mass and fat mass.
Physical functioning | baseline- 6 weeks -12 weeks- 6 months - 12 months post-diagnosis
  The PROMIS physical function short form (PROMIS-PF-SF) (questionnaire) will be used to measure physical functioning. It is composed of 10, 5-point Likert-scale items. A higher PROMIS T-score represents more of the concept being measured.
Radiotherapy-related fibrosis | baseline- 6 weeks -12 weeks
  Medical Research Council Rating Scale for Fibrosis: 4-point rating scale ranging from none to very marked density, retraction, and fixation.
Radiotherapy-related fibrosis | 6 months - 12 months
  RTOG Late Radiation Morbidity Scoring Scheme : 0-4 scale with descriptors for each category. Health provider administered, based on patient symptoms: 0 - absence of radiation effects, 5 - effects led to death. Severity of reaction is graded from 1-4.
Depression, anxiety, stress | baseline- 6 weeks -12 weeks- 6 months - 12 months post-diagnosis
  The Depression, Anxiety and Stress Scale-21 (DASS-21)(questionnaire) will be used. The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress.
  The rating scale is as follows: 0 Did not apply to me at all- 1 Applied to me to some degree, or some of the time - 2 Applied to me to a considerable degree or a good part of time - 3 Applied to me very much or most of the time.
  Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content.
Self-efficacy | baseline- 6 weeks -12 weeks- 6 months - 12 months post-diagnosis
  General Self-Efficacy Scale (questionnaire). This scale is a self-report measure of self-efficacy with 10 items (scored from 1-4). The total score is calculated by finding the sum of the all items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Stage of readiness to change | baseline -12 weeks
  The Physician-based Assessment and Counseling for Exercise (PACE) has 8 items intended to identify the patient's stage of readiness to begin a physical activity program.
Motivation towards exercise | baseline -12 weeks
  Behavioral Regulation in Exercise Questionnaire 2 will be used to assess motivation towards exercise. The BREQ-2 is a 19 item questionnaire that measures the stages of the self-determination continuum with respect to motivation to exercise with a 5 point Likert scale (0=not true for me, 4=very true for me)
Upper limb function | baseline- 6 weeks -12 weeks- 6 months - 12 months post-diagnosis
  The short version of the Disability of Arm, Shoulder and Hand - questionnaire will be used to evaluate upper limb function. The QuickDASH is a shortened version of the DASH Outcome Measure. Instead of 30 items, the QuickDASH uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb. The resultant score is reported on a scale of 0 to 100, where 0 represents no disability and 100 represents total disability
Physical activity level | baseline- 6 weeks -12 weeks- 6 months - 12 months post-diagnosis
  Both the International Physical Activity Questionnaire and daily step count (accelerometry) will be used to determine the physical activity level.
  The IPAQ is a 27-item self-reported measure of physical activity for use with individual adult patients aged 15 to 69 years old.
Social participation | baseline- 6 weeks -12 weeks- 6 months - 12 months post-diagnosis
  Impact on Participation and Autonomy Questionnaire : The IPA is a questionnaire that focuses on autonomy and participation of people with chronic conditions. The perceived participation scale consists of 31 items which are assessed using a 5 point rating scale (1=very good and 5=very poor) and the problem scale contains 8 items which are assessed using a 3 point rating scale (0=no problem and 2=severe problem). A participation score (range: 30-155) and a problem score (0-16) are produced by summing items in each scale.
Return to work | baseline - 6 weeks -12 weeks- 6 months - 12 months post-diagnosis
  The subjects will be asked to report their return to work
Health-related quality of life | baseline - 6 weeks -12 weeks- 12 months post-diagnosis
  Health-related quality of life will be measured with the European Organisation for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.

OTHER OUTCOMES:
Feasibility of the CSEP: participation | baseline
  •Acceptance of the invitation to participate (eligible patients vs participants)
Feasibility of the CSEP: compliance | baseline, 12 weeks and/or 6 months
  •Compliance and adherence to the intervention schedule (e.g. adherence to CSEP program, intervention attendance and engagement in scheduled sessions, prescribed frequency, intensity, time and type of exercise, ..)(collected using a diary)
Feasibility of the CSEP: sample characteristics | baseline, 12 weeks and/or 6 months
  •Sample characteristics (based on education level, age, self-efficacy, type of cancer, …) to identify subgroups of head and neck patients who participate, adhere best to the program and would benefit the most of it
Feasibility of the CSEP: retention of participants | 6 months
  •Retention of participants by estimating 6-month follow-up rates
Feasibility of the CSEP: satisfaction | 12 weeks and 6 months
  •Satisfaction with the intervention: participants will be asked to response on a 5-point scale from 1 (not at all satisfied/no) to 5 (very satisfied/definitely yes)
safety: reported health risks associated with the CSEP | baseline, 12 weeks and/or 6 months
  •Safety of the procedures in the intervention: Physical Activity Readiness- Questionnaire.
  The PAR-Q is a simple self-screening tool that is used to determine the safety or possible risks of exercising based on a subjects health history, current symptoms, and risk factors.
  All the questions are designed to help uncover any potential health risks associated with exercise.
Feasibility of the CSEP in daily clinical practice | baseline, 12 weeks and/or 6 months
  In a subgroup of participants, a qualitative study on the feasibility of the CSEP in daily clinical practice will be organized. All participants will be invited at baseline, 12 weeks and 6 months to participate in focus groups to discuss acceptability, expectations and satisfaction with the CSEP and maintenance program over time (baseline up to 6 months follow-up). During the focus group, a research assistant will ask a series of Likert-scale rated and open-ended questions related to the acceptability, expectations, and satisfaction of the exercise program. Fifteen patients (based on their willingness to participate in the focus group) will participate in 2-3 focus groups per time point. All raised issues will be considered and the exercise program will be modified accordingly.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Nuyts, Prof, Principal Investigator — UZ/KU Leuven
Locations (1):
- University Hospital Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Van Aperen K, Nuyts S, Devoogdt N, Troosters T, De Vrieze T, Gursen C, De Groef A. Cross-cultural adaptation, validity and reliability of the Dutch version of the Lymphedema Symptom Intensity and Distress Survey-Head and Neck version 2.0 (LSIDS-H&N v2.0) in head and neck cancer patients. Disabil Rehabil. 2025 Sep 7:1-16. doi: 10.1080/09638288.2025.2554945. Online ahead of print. PMID 40914813
- [Derived] Van Aperen K, De Groef A, Troosters T, Elshout P, Nuyts S. Feasibility of a comprehensive supervised exercise program during and after treatment of head and neck cancer: a mixed-methods study. Support Care Cancer. 2025 Jan 16;33(2):107. doi: 10.1007/s00520-024-09112-y. PMID 39820655
- [Derived] Van Aperen K, De Groef A, Devoogdt N, De Vrieze T, Troosters T, Bollen H, Nuyts S. EffEx-HN trial: study protocol for a randomized controlled trial on the EFFectiveness and feasibility of a comprehensive supervised EXercise program during radiotherapy in Head and Neck cancer patients on health-related quality of life. Trials. 2023 Apr 15;24(1):276. doi: 10.1186/s13063-023-07170-x. PMID 37061715